CLINICAL TRIAL: NCT06020859
Title: New MCE System for Detection of Gastric Lesions
Brief Title: MCE-new for Detection of Gastric Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MCE-new
Record Dates: First submitted 2023-07-25; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Capsule Endoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NaviEC-2000Pro Gastro Scan (Experimental): NaviEC-2000Pro Gastro Scan is a new mode of NaviEC-2000Pro
  Interventions: Device: undergo NaviEC-2000Pro Gastro Scan mode
- NaviEC-2000Pro Routine gastric examination (Experimental): NaviEC-2000Pro Routine gastric examination is a mode of NaviEC-2000Pro
  Interventions: Device: NaviEC-2000Pro Routine gastric examination
- NaviEC-1000 Routine gastric examination (Active Comparator): NaviEC-1000 Routine gastric examination is a mode of NaviEC-1000
  Interventions: Device: NaviEC-1000 Routine gastric examination

INTERVENTIONS:
Device: undergo NaviEC-2000Pro Gastro Scan mode — Patients undergo NaviEC-2000Pro Gastro Scan mode.
  Arms: NaviEC-2000Pro Gastro Scan
Device: NaviEC-2000Pro Routine gastric examination — Patients undergo NaviEC-2000Pro Routine gastric examination mode.
  Arms: NaviEC-2000Pro Routine gastric examination
Device: NaviEC-1000 Routine gastric examination — Patients undergo NaviEC-1000 Routine gastric examination mode.
  Arms: NaviEC-1000 Routine gastric examination

SUMMARY:
Clinical application of magnetically controlled capsule endoscopy : a prospective self-controlled trial

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness and safety of using a new MCE system for routine gastric examination and automatic scanning. This study is a prospective, self controlled clinical trail, which includes adult patients who plan to undergo MCE examination. Patients will undergo three different tests during the experiment: NaviEC-2000Pro Gastro Scan, NaviEC-2000Pro routine gastric examination, NaviEC-1000 routine gastric examination.

ELIGIBILITY:
Inclusion Criteria:

* underwent gastric examination;
* At least 18 years old；
* Be able to provide informed consent.

Exclusion Criteria:

* With swallowing obstruction or disorders;
* With known or suspected gastrointestinal obstruction, stenosis and fistula;
* Have no conditions for surgery or refuse to undergo any abdominal surgery;
* Be allergic to or have other known contraindication or intolerance to the drug used in the study;
* With pacemakers or other electronic devices such as electronic cochlear implants, implanted magnetic metal drug infusion pumps, neurostimulators, and magnetic metal foreign bodies;
* Women during pregnancy;
* Currently enrolled in another clinical trial of a drug or device;
* Other conditions determined by the investigator to be inappropriate for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
the degree of gastric mucosal visualization | 2 weeks
  The overall observational integrity of the gastric mucosa is based on the evaluation of the mucosal visualization of several key anatomical sites in the stomach: cardia, fundus, gastric body, gastric horn, gastric antrum and pylorus. The evaluation criteria for mucosal visualization of each site are: good : adequate observation, ≥90% of the gastric mucosa can be observed; fair : good observation, 70-90% of the gastric mucosa can be observed; poor : inadequate observation, <70% of the gastric mucosa can be observed.

SECONDARY OUTCOMES:
The time of gastric examination | 2 weeks
  The total time MCE required to complete the stomach examination
detection of lesions | 2 weeks
  The detection of gastric lesions by MCE
Equipment operation evaluation | 2 weeks
  Operation fluency is defined as the smooth response between operation and real-time capsule shooting. Stability is defined as the stable ability to control the capsule in a fixed position; Comfort is defined as the operator's operating comfort during examination. They were all rated on a scale of 1-5, with 1 being the worst and 5 the best
Safety Assessment | 2 weeks
  Number and incidence of device-related adverse events and serious adverse events

REFERENCES:
- [Background] Jiang X, Qian YY, Liu X, Pan J, Zou WB, Zhou W, Luo YY, Chen YZ, Li ZS, Liao Z. Impact of magnetic steering on gastric transit time of a capsule endoscopy (with video). Gastrointest Endosc. 2018 Oct;88(4):746-754. doi: 10.1016/j.gie.2018.06.031. Epub 2018 Jul 11. PMID 30005825
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503